CLINICAL TRIAL: NCT06982326
Title: Investigation of the Effects of Mental Fatigue on Physical Performance and Perceived Psychophysiological Reactions in Young Soccer Players: A Field Based Study
Brief Title: Mental Fatigue and Performance in Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ersan Arslan, Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UGaziosmanpasa-3
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Performance; Soccer; Mental Fatigue
Keywords: Neuromuscular control; Fatigue; Cognitive fatigue; Soccer performance
MeSH Terms: conditions — Mental Fatigue; Fatigue

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) Participants were strictly separated and think their intervention is the main intervention. The same was true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Fatigue (MF+) (Other): During the MF+ session, before each physical testing phase, participants completed a 30-min Colour Word Stroop task (CST) to trigger
  Interventions: Other: MF+
- Control (MF-) (Other): Control
  Interventions: Other: MF-

INTERVENTIONS:
Other: MF+ — During the MF+ session, before each physical testing phase, participants completed a 30-min Colour Word Stroop task (CST) to trigger MF. The paper-based version of the CST was completed in quiet rooms following the same protocol as in previous studies. This prolonged cognitive task was reported to require sustained attention and automatic response inhibition and effectively induced MF through cognitive manipulation. ThyIt had ben Four colour words (red, blue, green and yellow) were randomly printed and participants were asked to verbalise the colour of each word.
  Arms: Mental Fatigue (MF+)
Other: MF- — During the control session, before each physical testing phase, participants watched emotionally neutral documentaries for 30 min.
  Arms: Control (MF-)

SUMMARY:
The study employed a randomized, parallel-group, between-subjects design in which participants were assigned to either the MF+ or MF- condition and completed a single testing session accordingly. All test sessions were conducted on synthetic turf pitches and comprised three stages of testing, which included assessments of aerobic and anaerobic endurance, jumping, agility, and balance. During the familiarization session, players were briefed on the study procedures, practiced the main tasks, and became accustomed to the equipment and environment used during the intervention. During the MF+ session, prior to each physical testing stage, participants completed a 30-minute Color-word Stroop task (CST) to induce MF. To minimize external influence, players were not prompted or verbally encouraged during testing. Immediately, after each session, ratings of perceived exertion (RPE 6--20) were recorded using the category-level Borg scale (29), and enjoyment was assessed using the exercise enjoyment scale, a bipolar instrument consisting of eight items scored on a 1-7 Likert scale.

DETAILED DESCRIPTION:
The study employed a randomized, parallel-group, between-subjects design in which participants were assigned to either the MF+ or MF- condition and completed a single testing session accordingly. Players were recommended to sleep for at least 7-8 hours, refrain from exercising at moderate to high intensity, and avoid consuming alcoholic or caffeinated beverages during the 24 hours before the intervention. Indoor and outdoor temperatures (25-28°C) and humidity levels (35-40%) were kept consistent across all intervention sessions. All test sessions were conducted on synthetic turf pitches and comprised three stages of testing, which included assessments of aerobic and anaerobic endurance, jumping, agility, and balance. During the familiarization session, players were briefed on the study procedures, practiced the main tasks, and became accustomed to the equipment and environment used during the intervention. During the MF+ session, prior to each physical testing stage, participants completed a 30-minute Color-word Stroop task (CST) to induce MF. Four color words (red, blue, green, and yellow) were randomly printed, and participants were required to verbally name the color of each word. During the control (MF-) session, prior to each physical testing stage, participants watched emotionally neutral documentaries for 30 minutes. Each testing session began with a standardized 15-minute warm-up, consisting of 5 minutes of low- to moderate-intensity running followed by 10 minutes of upper- and lower-extremity-specific dynamic stretching, mobility exercises, and change-of-direction drills. To minimize external influence, players were not prompted or verbally encouraged during testing. Immediately, after each session, ratings of perceived exertion (RPE 6--20) were recorded using the category-level Borg scale, and enjoyment was assessed using the exercise enjoyment scale, a bipolar instrument consisting of eight items scored on a 1-7 Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male soccer players
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 14 years old
* Having a chronic disease
* Contraindications for exercise

Ages: 15 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Aerobic performance assessment | From baseline to the end of measurement at 1 day
  The test consisted of shuttle runs between two landmarks placed 20 metres apart, and athletes were required to complete a short active recovery period by running or walking within 10 seconds after each shuttle run. The testing protocol typically includes a standardised warm-up followed by progressive shuttle runs until exhaustion. The distance travelled or the level reached before exhaustion is used to measure performance. The test was carried out on an artificial turf field according to the recommended procedures.
Countermovement jump performance assessment | From baseline to the end of measurement at 1 day
  Countermovement jump tests with arms free (CMJf) tests were used to test the performance of the players in the vertical jump test. Each player's CMJf jump height was measured via Optojump photoelectric cells (Microgate, Bolzano, Italy). To ensure proper recovery and reduce fatigue, players were given a passive rest period of 2 minutes between consecutive trials in the same jump test. In addition, there was a rest period of 5 min between the different jump tests.
Agility performance assessment | From baseline to the end of measurement at 1 day
  Players completed three Zig-Zag agility tests with a ball (ZZwB) on a synthetic turf field. Each set was followed by a 3-minute recovery period, and the fastest time recorded from all sets was considered to be the performance of the test. The ZZwB trail comprises four 5-meter sections designed at 100° angles. In a previous study by Mirkov et al. (34), a coefficient of variation of 21.12%, intraclass correlation coefficients (ICCs) of 0.81 and 0.84, and typical measurement errors of 0.21 and 0.098 were reported for ZZwB.
Balence performance assessment | From baseline to the end of measurement at 1 day
  The Y balance test was used for balance measurements. Before the test, the length of both legs of each player was measured via a standard tape measure from the anterior superior iliac spine to the most distal medial malleolus in the supine position. The test, consisting of three different directions of movement (anterior, posteromedial, and posterolateral), was used to assess dynamic balance with a single-leg stance while reaching these directions. After six trials on each foot for familiarization, each player performed three successful reaches 15 s apart. After the test, the composite score (CS) was calculated via the following formula (37): CS = [(maximum anterior reach + maximum posteromedial reach + maximum posterolateral reach)/(leg length × 3)] × 100.
Anaerobic Endurance assessment | From baseline to the end of measurement at 1 day
  A three-corner run test (TCRT) was used to assess the speed and anaerobic endurance of the players. After the start signal, the players ran to a flagpole 80 m away from the start. The players then turned to the left side and ran to a flagpole, 20 m away from flagpole. After that, the players returned to flagpole 82.4 m from the start. Finally, turning to the right, the players ran to finish line and crossed the line to end the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa Universty, Tokat Province, Turkey, Turkey (Türkiye)

REFERENCES:
- [Background] Arslan E, Soylu Y, Clemente FM, Hazir T, Kin Isler A, Kilit B. Short-term effects of on-field combined core strength and small-sided games training on physical performance in young soccer players. Biol Sport. 2021 Oct;38(4):609-616. doi: 10.5114/biolsport.2021.102865. Epub 2021 Feb 11. PMID 34937971
- [Background] Soylu Y, Ramazanoglu F, Arslan E, Clemente FM. Effects of mental fatigue on the psychophysiological responses, kinematic profiles, and technical performance in different small-sided soccer games. Biol Sport. 2022 Oct;39(4):965-972. doi: 10.5114/biolsport.2022.110746. Epub 2021 Dec 30. PMID 36247954